CLINICAL TRIAL: NCT06061900
Title: Group Interval Fitness Program for Adolescents With Cognitive Impairments in the School Setting.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 23-0605
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Individuals completing pre and post-testing will be blinded to if the participate received the intervention or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants who receive group exercise intervention (Experimental): Intervention will include a warm-up, restive exercises with dumbbells, interval training, game or dancing, and cool down. Intervention sessions will run for 30-45 minutes, 2-3 times a week, for 8 weeks. Participants will also participate in pre and post-testing.
  Interventions: Other: Group exercise program
- Participants who do not receive group exercise intervention (No Intervention): Participants will participate in pre and post-testing.

INTERVENTIONS:
Other: Group exercise program — Group fitness program
  Arms: Participants who receive group exercise intervention

SUMMARY:
This study examines the outcomes of a group interval fitness program for secondary students with cognitive impairments in the school setting. It is well documented in the literature that individuals with cognitive impairments and medical conditions are at an increased risk for a sedentary lifestyle, obesity, and poor health-related fitness. These factors may further contribute to difficulties with planning for transitions from high school to young adulthood, independent or supported employment, and functional activities of daily living. An eight-week resistive exercise program was designed for secondary students with significant cognitive impairments who are participating in physical education classes as part of their standard curriculum. The goal of this study is to compare the outcomes related to strength, mobility, and functional activities for students in the intervention group compared to students who do not participate in this group interval program. This study investigates several important questions. Is a group fitness program effective in a school-based setting? Do individuals with cognitive impairments benefit from a group fitness program? Can a group fitness program correlate to functional and/or participation changes? With a group fitness program can changes be seen in lower extremity strength, upper extremity strength, grip strength, and mobility? How does a structured exercise group compare to a physical education class? Do physical education classes provide enough intensity for students with cognitive impairments?

DETAILED DESCRIPTION:
This prospective cohort study will compare students who received an exercise intervention group to those who did not. The cohorts share some things in common such as IQ, ambulatory status, and attending a physical education class.

Intervention will include a warm-up, restive exercises with dumbbells, interval training, game or dancing, and cool down. Intervention sessions will run for 30-45 minutes, 2-3 times a week, for 8 weeks.

Warm-up - 2-5 minutes

Dumbbells - 10-15 minutes

Interval training - 10-15 minutes

Game/Dance/Cool Down - 10 minutes

Pre and post-testing will be completed by a trained physical therapist, occupational therapist, or student of physical therapy who is completing a supervised clinical internship under a licensed physical therapist. Prior to any testing, the PI will conduct training sessions to ensure consistency between all testers. Pre and post-testing will be completed by a different group of physical therapists, occupational therapists, or students of physical therapy than the individuals providing the intervention. Individuals leading the intervention sessions will attend training sessions on the protocol and could be a physical therapist, occupational therapist, student physical therapist, adapted physical education teacher, or teacher.

High school and middle school buildings will be assigned into two groups: control and intervention, with the goal to have 5-6 buildings in each group. Participants in the control buildings will participate in pre and post-testing at the start and end of the eight-week program. During the eight weeks, participants in control buildings will continue with their normally scheduled physical education classes. Participants in the intervention buildings will also complete pre and post-testing and attend the fitness program during the eight weeks. Participants in the intervention buildings will attend their regularly scheduled physical education classes 2-3 times a week and the intervention group fitness program the other 2-3 days.

ELIGIBILITY:
Inclusion Criteria:

1. Must be enrolled in a secondary school within the Aurora Public Schools district and attend a physical education class.
2. Cognitive IQ less than 70 on a standardized measure documented in an Individualized Education Plan or Evaluation.
3. Ambulatory without an assistive device.
4. Not receiving intensive Physical Therapy services during the study or prior six months.
5. Able to follow verbal instructions for completing exercises, physical activities, and outcome measures.
6. At the time of the study, the participant does not have any acute orthopedic injuries that would impact active participation in physical education.

   -

Exclusion Criteria:

1. Student is unable to follow verbal instructions for completing exercise, physical activities, and outcome measures.
2. Student is 18 years old.
3. Student used a wheelchair or assistive device for primary mobility.

   -

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-10-23 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Test | 6 minutes
  The 6MWT measures the distance an individual can walk in six minutes on a level, flat surface. Individuals are asked to walk as fast as possible without running or being unsafe. This test is a submaximal exercise test used to measure function and endurance.

SECONDARY OUTCOMES:
Functional Strength Tests | 30 second intervals
  FST is comprised of three individual subtests including 30 seconds sit to stand, 30 seconds lateral step ups, and 30 seconds half-kneel to stand. Both half-kneel to stand and lateral step ups are completed on each leg. The individual is asked to complete as many repetitions as possible within the 30 second time frame. These tests measure lower extremity strength in a functional manner.

CONTACTS AND LOCATIONS:
Overall Officials: Holly L Ingham, DPT, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wouters M, Evenhuis HM, Hilgenkamp TIM. Physical fitness of children and adolescents with moderate to severe intellectual disabilities. Disabil Rehabil. 2020 Sep;42(18):2542-2552. doi: 10.1080/09638288.2019.1573932. Epub 2019 Apr 11. PMID 30973765
- [Result] Wang A, Gao Y, Wang J, Brown TJ, Sun Y, Yu S, Tong TK, Zhong LLD, Fong SSM, Dutheil F, Baker JS. Interventions for health-related physical fitness and overweight and obesity in children with intellectual disability: Systematic review and meta-analysis. J Appl Res Intellect Disabil. 2022 Sep;35(5):1073-1087. doi: 10.1111/jar.12999. Epub 2022 Apr 20. PMID 35445495
- [Result] Oppewal A, Hilgenkamp TI, van Wijck R, Schoufour JD, Evenhuis HM. Physical fitness is predictive for a decline in the ability to perform instrumental activities of daily living in older adults with intellectual disabilities: Results of the HA-ID study. Res Dev Disabil. 2015 Jun-Jul;41-42:76-85. doi: 10.1016/j.ridd.2015.05.002. Epub 2015 Jun 14. PMID 26079525
- [Result] Yuksel HS, Sahin FN, Maksimovic N, Drid P, Bianco A. School-Based Intervention Programs for Preventing Obesity and Promoting Physical Activity and Fitness: A Systematic Review. Int J Environ Res Public Health. 2020 Jan 3;17(1):347. doi: 10.3390/ijerph17010347. PMID 31947891
- [Result] Collins K, Staples K. The role of physical activity in improving physical fitness in children with intellectual and developmental disabilities. Res Dev Disabil. 2017 Oct;69:49-60. doi: 10.1016/j.ridd.2017.07.020. PMID 28818714